CLINICAL TRIAL: NCT02267902
Title: A Phase I, Open-Label, 2-Part Microtracer Study to Establish Absolute Bioavailability and the Absorption, Metabolism and Excretion of DA-1229 in Healthy Male Subjects
Brief Title: Microtracer Study to Establish Absolute Bioavailability and the Absorption, Metabolism, Excretion of DA-1229
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DA1229_BAMB_I
Record Dates: First submitted 2014-10-13; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

ARMS (2):
- Part 1 (Experimental): Single oral therapeutic dose of 5mg DA-1229 as a tablet + An IV dose of 20㎍ [14C]-DA-1229
  Interventions: Drug: DA-1229
- Part 2 (Experimental): Single oral therapeutic dose of 5mg [14C]-DA-1229
  Interventions: Drug: DA-1229

INTERVENTIONS:
Drug: DA-1229

SUMMARY:
The objectives of this study are to evaluate the absolute bioavailability, and absorption and excretion of DA-1229, an IMP in clinical assessment for the treatment of T2DM. The oral and IV PK of DA-1229 will also be evaluated. The metabolism of DA-1229 may also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 18 to 55
* BMI 18.0 to 30.0 kg/㎡

Exclusion Criteria:

* History of any drug or alcohol abuse in the past 2years
* Regular alcohol consumption nin males >21 units per week
* Current smokers and those who have smoked within the last 12months
* Radiation Exposure
* Positive drugs of abuse test result
* Positive HBsAg, HCV Ab, HIV results
* Serious adverse reaction or hypersensitivity to any drug of the formulation excipients
* Clinically significant allergy
* Donation of loss of blood within the previous 3 months
* Taking any prescribed or OTC drug or herbal remedies in the 14days before IMP administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
the absolute bioavailability of DA-1229 (F) | 240 hours
The mass balance recovery (Ae, %Ae) | 240 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Nottingham, Ruddington, United Kingdom